CLINICAL TRIAL: NCT05774483
Title: Sentinel Node Biopsy Versus Limited Elective Neck Dissection in Early Cancers of Oral Cavity NoDe Negative (SECOND N0): Non-inferiority Phase III Trial
Brief Title: Sentinel Node Biopsy Versus Limited Elective Neck Dissection in Early Cancers of Oral Cavity NoDe Negative
Acronym: SECOND N0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Richa Vaish, Professor and Surgeon, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4081
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-10

CONDITIONS: Mouth Neoplasms; Oral Cancers; Oral Squamous Cell Carcinoma (OSCC); Oral Squamous Cell Carcinomas; Sentinel Lymph Node Biopsy; Sentinel Lymph Node Biopsy (SLNB); Sentinel Lymph Node
Keywords: mouth neoplasms; neck dissection; sentinel lymph node biopsy; survival; morbidity; oral cancers; oral squamous cell carcinoma
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sentinel node biopsy (Active Comparator)
  Interventions: Procedure: Sentinel Node Biopsy
- Limited elective neck dissection (Experimental)
  Interventions: Procedure: Limited Elective Neck Dissection

INTERVENTIONS:
Procedure: Sentinel Node Biopsy — The Sentinel node will be localized after injecting peritumoral nano colloid followed by dynamic lymphoscintigraphy and SPECT localization. Methylene blue or indocyanine green may be used but not mandatory as an adjunct for lymphoscintigraphy for node localization. Intraoperatively the node will be identified using a hand-held gamma probe. The sentinel node will be processed on a frozen section, histopathological processing with serial step sectioning, and immunohistochemistry. If reported as metastatic, then a single-stage or second-stage completion neck dissection will be performed.
  Arms: Sentinel node biopsy
Procedure: Limited Elective Neck Dissection — Patients who are allocated to the limited END arm will undergo dissection of level I, IIa and III/IV nodes sparing level IIb. Level IIa will be subjected to a frozen section and if reported as metastatic will mandate clearance of level IIb.
  Arms: Limited elective neck dissection

SUMMARY:
The goal of this clinical trial is to compare the survival outcomes, morbidity and cost-effectiveness of sentinel node biopsy versus limited elective neck dissection in node-negative early oral cancers.

The main questions it aims to answer are:

* Survival outcomes
* Morbidity outcomes
* Cost-effectiveness

Participants will either undergo sentinel node biopsy followed by completion neck dissection if sentinel node is reported to be metastatic (SNB) or limited elective neck dissection where level IIb will be cleared only if level IIa is metastatic (limited END). The study will compare the outcomes in the two cohorts.

DETAILED DESCRIPTION:
Based on the current literature, we know that elective neck dissection (END) is mandatory in clinically node-negative early oral cancers. However, this leads to overtreatment and morbidity in about 55-80% of patients. The emergence of recent level I evidence makes SNB the standard of care in this setting. However, its limitation of being a two-staged procedure, steep learning curve, the burden on resources, lack of infrastructure, short-lasting decrease in morbidity and lack of cost-effectiveness data limits its wide applicability. It is our routine departmental practice of performing limited neck dissection clearing level I-III/IV sparing level IIb which is cleared only if level IIa is metastatic. It is hypothesized that limited END would limit the morbidity of shoulder dysfunction and be a more feasible and cost-effective treatment option which could be a suitable alternative to SNB in this setting without compromising the survival outcomes. With this background, we propose to embark upon a phase III RCT comparing the oncologic outcomes and morbidity of SNB versus limited END. We hypothesize that limited END would have survival outcomes non-inferior, morbidity similar to SNB with higher cost-effectiveness.

Aims and objectives:

Aim To compare the survival outcomes, morbidity and cost-effectiveness of SNB versus limited END in node-negative early oral cancers

Primary objective

1) Overall survival

Secondary objectives

1. Shoulder morbidity (key secondary endpoint) longitudinally up to 2 years
2. Disease-free survival
3. Neck nodal recurrence-free survival
4. Other side effects (chyle leak, hematoma, lymphoedema)
5. Longitudinal Quality of life up to 2 years
6. Cost-effective analysis

Exploratory objectives Blood and tumour tissue will be collected and banked for biomarker studies. Exploratory analyses will be conducted at a later date. Efforts may be directed to identify the biomarkers to predict nodal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Biopsy-proven invasive squamous cell carcinoma involving the site tongue and buccal mucosa
3. T1 and T2 lesions as per AJCC TNM 8 edition
4. Clinicoradiologically node negative
5. Amenable to per oral excision
6. Treatment naïve
7. No other site of malignancy

Exclusion Criteria:

1. Previous surgery in the head and neck region,
2. Upper alveolar or palatal lesions
3. Large heterogeneous leukoplakia or other premalignant lesions
4. Previous malignancy in the head and neck region
5. Patients requiring the free flap reconstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Defined from the date of randomization to death due to any cause

SECONDARY OUTCOMES:
Shoulder morbidity | Longitudinally at preoperatively, 3 months, at 6 months, 12 months and 24 months of treatment
  It will be assessed using the neck dissection impairment index (NDII). The range of movement of the shoulder will also be assessed using a goniometer
Neck nodal recurrence | 3 years
  Defined from the date of randomization to isolated neck node recurrence or death due to any cause
Disease free survival | 3 years
  Defined from the date of randomization to any recurrence (local, regional or distant metastasis) and second primary in the oral cavity
Health related Quality of life | Longitudinally at preoperatively, 3 months, at 6 months, 12 months and 24 months of treatment
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ C30 and QLQ HN35 instruments
Adverse events related to the surgical procedure and lymphedema | The lymphedema rating will be done at 3 months, at 6 months, 12 months and 24 months of treatment
  Details of the intra and perioperative delay including injury to critical structures, chyle leak, haemorrhage, and head and neck lymphedema
Cost effectiveness | 3 years
  Based on direct cost comparison

CONTACTS AND LOCATIONS:
Overall Officials: Richa Vaish, MS, M.Ch, Principal Investigator — Tata Memorial Hospital
Locations (3):
- India (3):
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - ACTREC, Navi Mumbai, Maharashtra
  - Mpmmcc & Hbch, Varanasi, Uttar Pradesh

REFERENCES:
- [Background] Garrel R, Poissonnet G, Moya Plana A, Fakhry N, Dolivet G, Lallemant B, Sarini J, Vergez S, Guelfucci B, Choussy O, Bastit V, Richard F, Costes V, Landais P, Perriard F, Daures JP, de Verbizier D, Favier V, de Boutray M. Equivalence Randomized Trial to Compare Treatment on the Basis of Sentinel Node Biopsy Versus Neck Node Dissection in Operable T1-T2N0 Oral and Oropharyngeal Cancer. J Clin Oncol. 2020 Dec 1;38(34):4010-4018. doi: 10.1200/JCO.20.01661. Epub 2020 Oct 14. PMID 33052754
- [Background] D'Cruz AK, Vaish R, Kapre N, Dandekar M, Gupta S, Hawaldar R, Agarwal JP, Pantvaidya G, Chaukar D, Deshmukh A, Kane S, Arya S, Ghosh-Laskar S, Chaturvedi P, Pai P, Nair S, Nair D, Badwe R; Head and Neck Disease Management Group. Elective versus Therapeutic Neck Dissection in Node-Negative Oral Cancer. N Engl J Med. 2015 Aug 6;373(6):521-9. doi: 10.1056/NEJMoa1506007. Epub 2015 May 31. PMID 26027881
- [Background] Hutchison IL, Ridout F, Cheung SMY, Shah N, Hardee P, Surwald C, Thiruchelvam J, Cheng L, Mellor TK, Brennan PA, Baldwin AJ, Shaw RJ, Halfpenny W, Danford M, Whitley S, Smith G, Bailey MW, Woodwards B, Patel M, McManners J, Chan CH, Burns A, Praveen P, Camilleri AC, Avery C, Putnam G, Jones K, Webster K, Smith WP, Edge C, McVicar I, Grew N, Hislop S, Kalavrezos N, Martin IC, Hackshaw A. Nationwide randomised trial evaluating elective neck dissection for early stage oral cancer (SEND study) with meta-analysis and concurrent real-world cohort. Br J Cancer. 2019 Nov;121(10):827-836. doi: 10.1038/s41416-019-0587-2. Epub 2019 Oct 15. PMID 31611612
- [Background] Dhar H, Vaish R, D'Cruz AK. Comment on "Nationwide randomised trial evaluating elective neck dissection for early-stage oral cancer (SEND study) with meta-analysis and concurrent real-world cohort.". Br J Cancer. 2020 Sep;123(7):1198-1199. doi: 10.1038/s41416-020-0981-9. Epub 2020 Jul 16. No abstract available. PMID 32669674
- [Background] Vaish R, Hawaldar R, Gupta S, Dandekar M, Shah S, Chaukar D, Pantvaidya G, Deshmukh A, Chaturvedi P, Pai P, Nair D, Nair S, Thakur M, Ghosh-Laskar S, Agarwal JP, D'Cruz AK. N0 neck trial: Does intensification of follow-up (Ultrasound + Physical Examination) influence outcomes in early-stage oral cancer? Eur J Cancer. 2024 Jun;204:114064. doi: 10.1016/j.ejca.2024.114064. Epub 2024 Apr 16. PMID 38705028